CLINICAL TRIAL: NCT05761223
Title: A Phase I/II, Open-label Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of FB849 Administered in Subjects With Advanced Solid Tumors Alone and in Combination With Pembrolizumab
Brief Title: A Phase I/II, Open-label Study to Investigate the Safety, Tolerability, PK, and Preliminary Efficacy of FB849
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: 1ST Biotherapeutics, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FB849_P101; KEYNOTE-F25 (Other: Merck Sharp & Dohme LLC); MK-3475-F25 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2023-02-20; First posted 2023-03-09 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: The study will be conducted in 3 parts: Phase I dose-escalation part with FB849 monotherapy and Phase II dose-escalation and dose-expansion parts of FB849 in combination with pembrolizumab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Phase Ia dose-escalation part of FB849 Monotherapy (Experimental): Participations will receive FB849 orally once a day.
  Interventions: Drug: Phase Ia dose-escalation part of FB849 Monotherapy
- Phase Ib dose-expansion of FB849 monotherapy (Experimental): Participations will receive FB849 orally once a day.
  Interventions: Drug: Phase Ib dose-expansion of FB849 monotherapy
- Phase IIa dose-escalation part of FB849 in Combination with Pembrolizumab (Experimental): Participations will receive FB849 orally once a day in combination with pembrolizumab.
  Interventions: Drug: Phase IIb dose-escalation part of FB849 in Combination with Pembrolizumab
- Phase IIb dose-expansion part of FB849 in Combination with Pembrolizumab (Type A cancer) (Experimental): Participations will receive FB849 orally once a day in combination with pembrolizumab.
  Interventions: Drug: Phase IIb dose-expansion part of FB849 in Combination with Pembrolizumab (Type A cancer)
- Phase IIb dose-expansion part of FB849 in Combination with Pembrolizumab (Type B cancer) (Experimental): Participations will receive FB849 orally once a day in combination with pembrolizumab.
  Interventions: Drug: Phase IIb dose-expansion part of FB849 in Combination with Pembrolizumab (Type B cancer)
- Phase IIb dose-expansion part of FB849 in Combination with Pembrolizumab (Type C cancer) (Experimental): Participations will receive FB849 orally once a day in combination with pembrolizumab.
  Interventions: Drug: Phase IIb dose-expansion part of FB849 in Combination with Pembrolizumab (Type C cancer)

INTERVENTIONS:
Drug: Phase Ia dose-escalation part of FB849 Monotherapy — At a given level dose once daily
  Other Names: FB849
  Arms: Phase Ia dose-escalation part of FB849 Monotherapy
Drug: Phase Ib dose-expansion of FB849 monotherapy — At recommended dose for expansion cohort once daily
  Other Names: FB849
  Arms: Phase Ib dose-expansion of FB849 monotherapy
Drug: Phase IIb dose-escalation part of FB849 in Combination with Pembrolizumab — At recommended dose for expansion cohort once daily in combination with pembrolizumab
  Other Names: FB849; KEYTRUDA®
  Arms: Phase IIa dose-escalation part of FB849 in Combination with Pembrolizumab
Drug: Phase IIb dose-expansion part of FB849 in Combination with Pembrolizumab (Type A cancer) — At recommended dose for expansion cohort once daily in combination with pembrolizumab
  Other Names: FB849; KEYTRUDA®
  Arms: Phase IIb dose-expansion part of FB849 in Combination with Pembrolizumab (Type A cancer)
Drug: Phase IIb dose-expansion part of FB849 in Combination with Pembrolizumab (Type B cancer) — At recommended dose for expansion cohort once daily in combination with pembrolizumab
  Other Names: FB849; KEYTRUDA®
  Arms: Phase IIb dose-expansion part of FB849 in Combination with Pembrolizumab (Type B cancer)
Drug: Phase IIb dose-expansion part of FB849 in Combination with Pembrolizumab (Type C cancer) — At recommended dose for expansion cohort once daily in combination with pembrolizumab
  Other Names: FB849; KEYTRUDA®
  Arms: Phase IIb dose-expansion part of FB849 in Combination with Pembrolizumab (Type C cancer)

SUMMARY:
This is the first-in-human, multicenter, open-label Phase I/II study to investigate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and preliminary efficacy of FB849 alone and in combination with pembrolizumab in subjects with advanced solid tumors for whom no standard therapy is available.

DETAILED DESCRIPTION:
The study will be conducted in 3 parts: Phase I dose-escalation part with FB849 monotherapy and Phase II dose-escalation and dose-expansion parts of FB849 in combination with pembrolizumab.

The Phase Ia dose-escalation part will use an adaptive study design termed Bayesian optimal interval (BOIN) design to investigate the safety and tolerability of FB849, and determine the maximum tolerated dose (MTD) and preliminary recommended Phase II dose (RP2D) of FB849. A BOIN design is a hybrid of rule-based and model-based design, which has the flexibility of dose escalation and de-escalation and allows more subjects to be enrolled into the doses closest to the target toxicity rate.

Phase IIa enrollment will be initiated after Stage 1 of Phase Ib is completed. The selected RP2D from the prior Phase Ib part and a dose level ≥ 1 dose lower than the RP2D of FB849 will be selected by the SMC and will be evaluated in combination with a standard dose of pembrolizumab. Dose escalation will follow a BOIN design, but with at least 6 subjects at each FB849 dose level.

In the Phase IIb part of the study, subjects with Type A cancer, Type B cancer, or Type C cancer will be enrolled in 3 cohorts to evaluate FB849 at the RP2D in combination with a standard dose of pembrolizumab to provide assessments of safety and anti-tumor activity of FB849. Both Phase II parts will also explore the impact of FB849 on pharmacodynamics and metabolites when in combination with pembrolizumab. Enrollment to Phase IIb will follow a Simon's two -stage design enrollment.

Subjects will be monitored for safety, tolerability, and preliminary efficacy throughout the study. Tumor response will be assessed by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 approximately every 6 weeks (± 3 days) in the first 18 weeks, then every 9 weeks (± 7 days) thereafter until disease progression, using computed tomography or magnetic resonance imaging of the chest, abdomen/pelvis, and if clinically indicated additional assessments eg, craniocerebral imaging, bone scan. Treatment with FB849 will continue until the start of a new anti-cancer treatment, disease progression, subject refusal, unacceptable toxicity, death, lost to follow-up, etc, whichever occurs first. Subjects who discontinue treatment due to other reasons than disease progression will continue with tumor assessments as per protocol until disease progression, death, or starting a new anti-cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject should understand, sign, and date the written ICF prior to screening.
* Male or female aged 18 years or older.
* Subjects must have at least 1 measurable target lesion according to RECIST version 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Life expectancy ≥ 3 months in the opinion of the investigator.
* Adequate organ function and bone marrow function as indicated by the following screening assessments performed within 14 days prior to the first dose of study treatment

Exclusion Criteria:

* Known allergy or hypersensitivity to any component of the study treatment.
* Has a known additional malignancy that is progressing or has required active treatment.
* Has abnormal or inadequately controlled endocrine function.
* Inability to take oral medication or significant nausea and vomiting, malabsorption, external biliary shunt, or significant bowel resection that would preclude adequate absorption of oral medication.
* Previous anti-cancer therapy, including chemotherapy (chemotherapy with nitrosourea or mitomycin should be at least 6 weeks prior to initiation of study treatment), radiotherapy, molecular targeted therapy, or other investigational drugs received ≤ 4 weeks; endocrine therapy ≤ 2 weeks or ≤ 5-half-lives (whichever is shorter) prior to initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of FB849 and to identify maximum tolerated dose (MTD)/ recommended Phase II dose (RP2D) and dosing schedule of FB849 in subjects with advanced solid tumors | DLT Assessment at the end of Cycle 1(each cycle is 21 days.)
  The MTD is defined to be the highest safe dose with an estimated DLT rate less than 30.

SECONDARY OUTCOMES:
To determine the pharmacokinetic parameters such as Peak Plasma Concentration (Cmax) of FB849 | Blood: Predose, 1, 2, 4, 8, 12, 24 hours postdose at C1D1 and C1D21; predose and 4, 8, and 24 hours postdose at C1D8; predose at C1D15; and predose on C2D1, C4D1, and C6D1, Urine: predose and 0-4 hour, 4-8 hour, 8-12 hour, 12-24 hour post-dose
  The PK parameters should include, where appropriate, area under the concentration-time curve (AUC), maximum observed concentration (Cmax), time to maximum observed concentration (tmax), and apparent terminal elimination half-life (t1/2), apparent total body clearance (CL/F), apparent volume of distribution (Vz/F), Cmax at steady state (Css-max), minimum observed concentration at steady state (Css-min), AUC at steady state (AUCss), accumulation ratio (Rac), amount excretion (Ae), fraction excretion (Fe), renal clearance (CLR).
To assess preliminary anti-tumor activity of FB849 | every 6 weeks (± 3 days) in the first 18 weeks, then every 12 weeks (± 7 days) thereafter until disease progression assessed up to approximately 3 years
  Tumor response will be assessed by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 using computed tomography (CT) or magnetic resonance imaging (MRI) of the chest, abdomen/pelvis, and additional assessments (e.g., craniocerebral imaging, bone scan) based on clinical indications.

CONTACTS AND LOCATIONS:
Overall Officials: 1STBIO Chief Development Officer, Study Director — 1ST Biotherapeutics
Locations (5):
- United States (5):
  - Cleveland Clinic, Cleveland, Ohio
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - NEXT Oncology San Antonio, San Antonio, Texas
  - Next Oncology Virginia, Fairfax, Virginia
  - Summit Cancer Centers - Spokane Valley, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No